CLINICAL TRIAL: NCT00185120
Title: A Study on the Efficacy and Safety of Olmesartan Medoxomil and Its Combination With Hydrochlorothiazide Compared With an ACE Inhibitor and Its Combination With a Calcium Channel Blocker in Patients With Stage 2 Hypertension
Brief Title: Treatment of High Blood Pressure Using Olmesartan With Hydrochlorothiazide Compared to an ACE Inhibitor With a Calcium Channel Blocker
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 866-447
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Hypertension
Keywords: Hypertension; angiotensin receptor blocker; calcium channel blocker; angiotensin converting enzyme inhibitor hydroclorothiazide
MeSH Terms: conditions — Hypertension | interventions — Olmesartan Medoxomil; benazepril; Amlodipine

INTERVENTIONS:
Drug: Olmesartan medoxomil
Drug: Hydroclorothiazide
Drug: Benazepril
Drug: Amlodipine

SUMMARY:
A comparison of 2 different combinations of high blood pressure medications to treat hypertension

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Patients with high blood pressure

Exclusion Criteria:

* Hypertensive encephalopathy, stroke or transient ischemic attack within the past 6 months
* History of myocardial infarction, percutaneous transluminal coronary revascularization, coronary artery bypass graft, and/or unstable angina pectoris within the past 6 months
* Type 1 diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152
Dates: Start 2005-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure from the start of the study

SECONDARY OUTCOMES:
Change in diastolic blood pressure from the start of the study
Percent of patients who achieve target blood pressure goals

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Mobile, Alabama
  - Memorial Research Medical Center, Long Beach, California
  - National Research Institute, Los Angeles, California
  - Clinical Trials Research, Roseville, California
  - Apex Research Institute, Santa Ana, California
  - Orange County Research Center, Tustin, California
  - Westlake Medical Center, Westlake Village, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - The Greater Fort Lauderdale Heart Group Research, Fort Lauderdale, Florida
  - SFBC International, Miami, Florida
  - CLIRECO, Inc., Tamarac, Florida
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Heartland Research Associates, Wichita, Kansas
  - Androscoggin Cardiology Research, Auburn, Maine
  - Internal Medicine Associates of Charlotte, Charlotte, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Omega Medical Research, Warwick, Rhode Island
  - Volunteer Research Group, University of Tennessee Med. Ctr., Knoxville, Tennessee
  - Punzi Medical Center, Carrollton, Texas